CLINICAL TRIAL: NCT03078634
Title: The MANTRA Study: The Multi-disciplinary Treatment of Functional Gut Disorders Study
Brief Title: The Multi-disciplinary Treatment of Functional Gut Disorders Study
Acronym: MANTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Responsible Party: Principal Investigator, Chamara Basnayake, Gastroenterologist, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MANTRA
Record Dates: First submitted 2017-02-24; First posted 2017-03-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Irritable Bowel Syndrome; Functional Dyspepsia; Constipation - Functional; Faecal Incontinence; Functional Abdominal Pain Syndrome; Other Rome IV Functional Gastrointestinal Disorders
Keywords: Irritable bowel syndrome; Constipation; Functional dyspepsia; Multi-disciplinary treatment
MeSH Terms: conditions — Irritable Bowel Syndrome; Encopresis; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Disciplinary clinic (Active Comparator)
  Interventions: Other: Multi-disciplinary clinic model
- Standard Gastrointestinal clinic (Placebo Comparator)
  Interventions: Other: Standard outpatient care

INTERVENTIONS:
Other: Multi-disciplinary clinic model — Clinic model incorporating multiple disciplines for the treatment of functional gut disorders. Disciplines include: gastroenterologists, psychiatrists, psychologists, hypnotherapists, behavioural therapists and dieticians. End of clinic case conference involving clinical disciplines will also occur to coordinate care.
  Arms: Multi-Disciplinary clinic
Other: Standard outpatient care — Standard care provided in outpatient clinics staffed by GI doctors only
  Arms: Standard Gastrointestinal clinic

SUMMARY:
Randomised controlled trial comparing standard outpatient clinic treatment with multi-disciplinary clinic treatment for functional gastrointestinal disorders. Patients will be followed up to end of clinic treatment and 12 months beyond the end of treatment. Symptoms, quality of life, costs to the healthcare system and psychological outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Functional gastrointestinal disorder as defined by Rome IV

Exclusion Criteria:

* Diagnosed or suspicion of organic gastrointestinal disorder (ie Coeliac, IBD)
* Age <18 or >80
* Non-English speaking
* Patient's from outside of metropolitan Melbourne who cannot attend clinic visits
* Prominent eating disorder
* Chronic opioid dependence
* Medications which can explain functional gut symptoms
* Surgery of GI tract that can explain functional gut symptoms
* Major, non-GI, organ dysfunction
* Pregnancy
* Major Psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with global improvement in their condition. | Definition of discharge timepoint: Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first.
  Global improvement in their condition is defined as a response of either "slightly better" or "much better" to the question: "Compared with before I was first seen in clinic, I feel my gut condition is now:". The question is marked on a 5-point likert scale: Much worse, slightly worse, same, slightly better, much better.

SECONDARY OUTCOMES:
Proportion of subjects, with Irritable bowel syndrome or centrally mediated abdominal pain syndrome, with a 50% reduction in Irritable bowel syndrome severity scoring system (IBS-SSS) | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
Proportion of subjects with constipation who score a 50% reduction in Cleveland clinic constipation scoring system | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
Proportion of subjects with faecal incontinence who score a 50% reduction in St Mark's Incontinence score | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
Proportion of subjects with functional dyspepsia who score a 50% reduction in the symptom score of the Nepean dyspepsia index | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
Quality of life as measured by RAND SF-36 v1 | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
Quality of life as measured by Euro-QOL EQ-5D | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
  Scores from the EQ-5D will be compared between groups and QALY will be derived from EQ-5D.
Psychological wellbeing as measured by hospital anxiety and depression score (HADS) | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B)12 months after discharge.
Proportion of subjects with who answer yes to: In the past 7 days, have you had adequate relief of your gut condition? [YES/NO] | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
Somatisation as measured by somatic symptom scale-8 (SSS-8) | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
Cost to the healthcare system | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
  $AUD per patient cost to the Australian healthcare system.
Proportion of subjects with global improvement in their condition. | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
  Global improvement in their condition is defined as a response of either "slightly better" or "much better" to the question: "Compared with before I was first seen in clinic, I feel my gut condition is now:". The question is marked on a 5-point likert scale: Much worse, slightly worse, same, slightly better, much better.
Proportion of subjects with a 50% reduction in gastrointestinal symptom severity index score | A) Day 1 of being discharged from clinic, or 9 months after baseline visit, whichever occurs first. B) 12 months after discharge.
  Patients will complete a GISSI (Gastrointestinal symptom severity index) questionnaire at time of "discharge from clinic" and 12 months after "discharge from clinic". The score used will be specific to their symptom cluster.

CONTACTS AND LOCATIONS:
Overall Officials: Chamara Basnayake, MBBS, Principal Investigator — Gastroenterologist / PhD candidate
Locations (1):
- St Vincent's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basnayake C, Kamm MA, Stanley A, Wilson-O'Brien A, Burrell K, Lees-Trinca I, Khera A, Kantidakis J, Wong O, Fox K, Talley NJ, Liew D, Salzberg MR, Thompson AJ. Long-Term Outcome of Multidisciplinary Versus Standard Gastroenterologist Care for Functional Gastrointestinal Disorders: A Randomized Trial. Clin Gastroenterol Hepatol. 2022 Sep;20(9):2102-2111.e9. doi: 10.1016/j.cgh.2021.12.005. Epub 2021 Dec 9. PMID 34896645
- [Derived] Basnayake C, Kamm MA, Stanley A, Wilson-O'Brien A, Burrell K, Lees-Trinca I, Khera A, Kantidakis J, Wong O, Fox K, Talley NJ, Liew D, Salzberg MR, Thompson AJ. Standard gastroenterologist versus multidisciplinary treatment for functional gastrointestinal disorders (MANTRA): an open-label, single-centre, randomised controlled trial. Lancet Gastroenterol Hepatol. 2020 Oct;5(10):890-899. doi: 10.1016/S2468-1253(20)30215-6. Epub 2020 Jul 14. PMID 32679040
- [Derived] Basnayake C, Kamm MA, Salzberg M, Khera A, Liew D, Burrell K, Wilson-O'Brien A, Stanley A, Talley NJ, Thompson AJ. Defining Optimal Care for Functional Gut Disorders - Multi-Disciplinary Versus Standard Care: A Randomized Controlled Trial Protocol. Contemp Clin Trials. 2019 Sep;84:105828. doi: 10.1016/j.cct.2019.105828. Epub 2019 Aug 19. PMID 31437539